CLINICAL TRIAL: NCT00241852
Title: Family Approach to Managing Asthma in Early Teens
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jean-Marie Bruzzese, Associate Professor, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 333; R01HL079953 (NIH)
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral Intervention: Asthma: It's a Family Affair (Experimental): Separate student and parent intervention groups.
  Interventions: Behavioral: Asthma: It's a Family Affair!
- Behavioral Control Group (Active Comparator): Students and parents participate in an education only control group
  Interventions: Behavioral: Asthma and Stress Comparator

INTERVENTIONS:
Behavioral: Asthma: It's a Family Affair! — Intervention families will receive a comprehensive program with two complementary components: (1) a school-based intervention to empower middle school students to manage their asthma and (2) parent training to teach their caregivers childrearing skills that support the youth's growing autonomy and need to self-manage their disease. The student component is comprised of 6, 60 minute group workshops; the caregiver component consists of 5, 90-minute group workshops.
  Arms: Behavioral Intervention: Asthma: It's a Family Affair
Behavioral: Asthma and Stress Comparator — Caregivers assigned to the Asthma and Stress Comparator group will receive a single educational workshop focusing on the developmental changes adolescents experience, how these changes may cause stress, and ways to cope with stress. The children will also participate in a single school-based session on similar topics. Both caregivers and students will learn basic asthma facts.
  Arms: Behavioral Control Group

SUMMARY:
The purpose of this study is to test two asthma management programs: (a) a school-based curriculum to empower middle school students to manage their asthma and (b) a parent training curriculum to teach childrearing skills that support the youths' growing autonomy and need to self-manage their disease.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a public health problem with its prevalence and morbidity being significant in 11- to 14-year olds, particularly among ethnic minorities. Despite this, little has been done to intervene with this age group. This is surprising considering the success of asthma education programs for younger children. In addition, there are no reports of parenting training to help families manage asthma despite the significant influence parenting strategies have on the management of chronic illnesses.

DESIGN NARRATIVE:

The overall goal of this study is to test the efficacy of a program with two complementary components: (a) a school-based curriculum to empower middle school students to manage their asthma and (b) a parent training curriculum to teach childrearing skills that support the youths' growing autonomy and need to self-manage their disease. The specific aims are: (1) to implement screening to identify 6th - 8th grade students with persistent asthma; and (2) to provide health education and parent training to help children and parents manage asthma more effectively. The student program is based on Coping with Asthma at Home and at School, a successful program developed in Holland. The parent program is an adaptation of Thriving Teens, an effective parent training program developed by the investigators. Participants in this randomized control trial will be 384 children with asthma and their caregivers from 16 New York City public schools serving low-income, ethnic minorities. It is hypothesized that students randomized to the intervention will have, relative to controls, improvements in three primary outcomes: (1) reduced symptom severity; (2) improved quality of life; and (3) better asthma management skills. Also, when compared to controls, intervention students will show improvement in the following secondary outcomes: (4) urgent health care utilization; (5) days with activity restriction; and (6) parent-child interactions. Caregivers and children will complete comprehensive surveys assessing these outcomes at baseline, and immediately and 6- and 12-months after the intervention.

ELIGIBILITY:
Inclusion Criteria for Youth:

* Prior diagnosis of asthma from a medical provider
* Asthma symptoms an average of 3 times per month during the 12 months prior to study entry OR less frequent symptoms but having 1 or more urgent visits to a doctor/emergency room or hospitalization for asthma during the 12 months prior to study entry
* Use of prescribed asthma medication in the 12 months prior to study entry

Inclusion Criteria for Families:

* Child and participating parent must live together

Exclusion Criteria for Youth:

* Co-morbidity that might affect lung function, such as cystic fibrosis or sickle cell anemia
* Highly specialized developmental or learning needs (e.g., Down's syndrome, mental retardation, severe ADHD)
* Major psychiatric illness

Exclusion Criteria for Families:

* Foster parents and their children

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 392 (Actual)
Dates: Start 2005-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Symptom severity | baseline, immediate post-intervention and every 2 months thereafter up to and including 12-months post-intervention
quality of life | Baseline, and immediate, 6-months and 12-months post-intervention
asthma management skills | Baseline, and immediate, 6-months and 12-months post-intervention

SECONDARY OUTCOMES:
Urgent health care utilization | baseline, immediate post-intervention and every 2 months thereafter up to and including 12-months post-intervention
days with activity restriction | baseline, immediate post-intervention and every 2 months thereafter up to and including 12-months post-intervention
parent-child interactions | Baseline, and immediate, 6-months and 12-months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Bruzzese, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Bruzzese JM, Unikel L, Gallagher R, Evans D, Colland V. Feasibility and impact of a school-based intervention for families of urban adolescents with asthma: results from a randomized pilot trial. Fam Process. 2008 Mar;47(1):95-113. doi: 10.1111/j.1545-5300.2008.00241.x. PMID 18411832